CLINICAL TRIAL: NCT04889547
Title: Randomized Controlled Trial Assessing the Effect of Intraoperative Dexamethasone in the Management of Postoperative Analgesia and Stiffness After Distal Radius Fixation
Brief Title: Randomized Controlled Trial Assessing the Effect of Dexamethasone on Postoperative Function After Distal Radius Fixation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 21-0069
Record Dates: First submitted 2021-04-05; First posted 2021-05-17 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Experimental): Patient will receive intraoperative dexamethasone during distal radius open reduction and internal fixation
  Interventions: Drug: Dexamethasone
- No dexamethasone (Placebo Comparator): Patient will not receive intraoperative dexamethasone during distal radius open reduction and internal fixation
  Interventions: Other: No dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Intraoperative intravenous dexamethasone
  Arms: Dexamethasone
Other: No dexamethasone — No intraoperative intravenous dexamethasone
  Arms: No dexamethasone

SUMMARY:
The study is designed to assess the use of intraoperative dexamethasone on postoperative analgesia and stiffness after open reduction and internal fixation of distal radius fractures. The idea is that the dexamethasone will aid in reducing postoperative swelling which will then improve pain control as well as overall function.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Willingness to comply with study procedures and
* Male or female greater than 18 years old
* American Society of Anesthesia class I/II/III
* Ability to take oral medicine in order to assess opioid regimen postop
* Distal radius open reduction and internal fixation surgery with single incision and volar plate
* Ability to consent for and receive a preoperative upper extremity nerve block by anesthesia

Exclusion Criteria:

* Chronic opioid users
* Prescriptions for selective-serotonin reuptake inhibitors, gabapentin, duloxetine within 3 days of surgery
* History of diabetes and A1C > 8
* Systemic glucocorticoids within 1 month of study enrollment
* Inability to take ibuprofen or acetaminophen due to allergy or condition
* History of hepatitis
* Pregnancy or lactation
* Allergic to opioids
* Known allergic reactions to components of IV dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Patient rated wrist evaluation | 48 hours, 1 week, 2 weeks
  15-item questionnaire designed to measure wrist pain and disability in activities of daily living. PWRE will be assessed at multiple time point to assess for change in the score. The higher the score, the more function exhibited.

SECONDARY OUTCOMES:
Finger-to-palm distance | 48 hours, 1 week, 2 weeks
  Objective measure to quantify stiffness. This is measured by measuring the distance from the tip of the third finger to the palm during attempted creation of a fist. FTP will be measured at multiple time points to assess for change.
Visual analog scale | 48 hours, 1 week, 2 weeks
  Validated, subjective measure for pain. Measured on a 10 point scale, 0 being no pain and 10 being maximum pain. VAS will be evaluated at multiple time points to assess for change.
Total opioid consumption | 48 hours, 1 week, 2 weeks
  Measuring total opioid consumption postoperatively. This will be measured by self reported mechanism. Assessed at multiple time points to assess for change.

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Yes